CLINICAL TRIAL: NCT02054962
Title: Persistent Pain and Associated Functional Decline Among Elderly Experiencing Motor Vehicle Collision
Brief Title: Persistent Pain Among Elderly Experiencing Motor Vehicle Collision
Acronym: Elderly CRASH
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11-0172; K23AG038548 (NIH)
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2017-04

CONDITIONS: Persistent Pain After Injury; Functional Decline After Injury
Keywords: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva samples collected for participants 1-150. Saliva, whole blood DNA and RNA collected for participants 151-250
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elderly: The investigators intend to asses the effect of fear of movement, PTSD symptoms, and physical activity on persistent pain and functional decline.

SUMMARY:
Chronic problems after traumatic events are common in non-elderly adults. Previous studies have shown that after minor motor vehicle collision (MVC), 10-30% of non-elderly adult patients develop chronic regional pain (neck or back pain). In addition, up to 1/3 of non-elderly adults will develop psychological sequelae, including posttraumatic stress disorder, depression, and anxiety disorders. There have been no prospective studies examining the frequency or predictors of persistent pain or psychological sequelae in older adults. The proposed study seeks to determine the frequency of persistent pain, psychological sequelae, and associated disability in older adults after minor MVC trauma and to identify candidate predictors for a model of adverse outcomes after MVC in this population. 200 individuals over 65 years of age will be recruited from emergency departments in four states with no-fault accident laws. Patients who meet inclusion criteria and who consent to the emergency department (ED) study will undergo a 30-45 minute ED assessment of crash-related, psychosocial, and biological factors, and complete telephone follow-ups at 2 weeks, 6 weeks 6 months, and 12 months. The wealth of information gained from this study will be used to determine the frequency of adverse events in older adults after MVC and to identify high risk elderly patients. These results will inform subsequent development of secondary pharmacologic and/or behavioral interventions to prevent chronic pain and psychological sequelae after traumatic events in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Patient speaks English, presented to ER less than 24 hours after an MVC, patient has an address and telephone

Exclusion Criteria:

* Patient
* is a prisoner,
* has fractures or an intracranial injury,
* has injuries that are life threatening or expected to result in hospitalization for more than 72 hours,
* is receiving end of life, hospice, or comfort care, or
* is considered ineligible by treating physician.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly experiencing motor vehicle collision
Sampling Method: Non-Probability Sample
Enrollment: 211 (Actual)
Dates: Start 2012-06; Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Average pain 6 months after Emergency Department visit | 6 months
  Average pain during the past week with pain measured on a 0-10 scale.

SECONDARY OUTCOMES:
Physical function at 6 months after Emergency Department visit | 6 months
  Function measured on a 0-12 scale based on patient reported ability or difficulty walking, carrying objects, and climbing stairs (Simonsick E, et al. 2001).

CONTACTS AND LOCATIONS:
Overall Officials: Timothy F Platts-Mills, MD, MSc, Study Director — UNC Chapel Hill
Locations (1):
- Spectrum Health - Butterworth Hospital, Grand Rapids, Michigan, United States